CLINICAL TRIAL: NCT06475924
Title: Relation Between Position of the Uterus (Anteversion or Retroversion Flexion) and Degree of Cesarean Scar Niche : Cross -Sectional Study
Brief Title: Relation Between Position of the Uterus (Anteversion or Retroversion Flexion) and Degree of Cesarean Scar Niche
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maya Abdelrazek, dr_maya89@med.asu.edu.eg, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS 522/2023
Record Dates: First submitted 2024-06-16; First posted 2024-06-26 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Anteversion of Uterus; Retroflex Uterus; CSD
Keywords: Cesarean scar defefect; Isthmocele; Caesarean scar niche; Anteverted uterus; Retroverted uterus
MeSH Terms: conditions — Uterine Retroversion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cesarean Scar Defect (CSD) (Other): cesarean scar niche/defect (CSD) by transvaginal ultrasound that is defined as "indentation at the site in the cesarean section scar with a depth of at least 2 mm" that was agreed upon in 2019 by a European task force
  Interventions: Diagnostic Test: Caesarean scar defect evlauation by ultraosund

INTERVENTIONS:
Diagnostic Test: Caesarean scar defect evlauation by ultraosund — Women will be examined in the lithotomy position with an empty bladder. The uterus will be examined in a standardized way excluding causes of abnormal uterine bleeding or pelvic pain (myoma, polyp, pelvic inflammatory disease, adenomyosis).
  Upon detection of the SCD, the following will be measured:
  In the midsagittal plane: the depth (the vertical distance between the base and apex of the defect), width (the length of the widest gap along the cervicoisthmic canal), residual myometrial thickness (RMT) overlying the defect, and the adjacent myometrial thickness fundal to the defect.
  In the transverse plane: the length of the defect.
  The uterine position will be classified as anteverted or retroverted.
  Clinical symptoms of the patients will be reviewed such as :Postmenstrual spotting, Abnormal uterine bleeding, Pain, Secondary infertility.

SUMMARY:
This study aims to determine the association between the size of caesarean scar niche and uterine position in childbearing women.

Research hypothesis: There is a relation between uterine position and degree of cesarean scar niche.

Research question: Is there a relation between uterine position and degree of cesarean scar niche?

DETAILED DESCRIPTION:
It has been noted that the cesarean scar defect in patients with retroflexed uteri appear to be larger than are those in patients with anteverted uteri.

This study will describe the association between position of the uterus whether share in degree of cesarean scar niche or not and associated symptoms.

Primary outcome:

The association between the position of the uterus (Anteverted/Retroverted) and large CSD (the ratio between the depth and adjacent myometrial thickness)

Secondary outcomes:

The association between position of the uterus (Anteverted/Retroverted) and:

* Residual myometrial thickness (RMT).
* Depth, Width, Length of SCD.

The association to the clinical symptoms as:

* Postmenstrual spotting: more than 2 days of intermenstrual spotting, or more than 2 days of brownish discharge after the end of menstruation if bleeding duration exceeds 7 days (discharge is considered normal if bleeding duration is < 7 days).
* Abnormal uterine bleeding (AUB) as per FIGO guideline.
* Pain as dysmenorrhea, chronic pelvic pain or dyspareunia. If present will be assed using Visual Analogue Scale (VAS).
* Secondary infertility: inability of a couple to conceive after one year of regular, unprotected intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Women in childbearing age.
* At least six months postpartum.
* With cesarean scar niche/defect (CSD) by transvaginal ultrasound that is defined as "indentation at the site in the cesarean section scar with a depth of at least 2 mm" that was agreed upon in 2019 by a European task force

Exclusion Criteria:

* Severely Obese (Body mass index; BMI more than or equal to 35 kg/m2).
* Women with abnormal uterine pathology, observed during the ultrasound examination that may have been responsible for abnormal uterine bleeding, including endometrial hyperplasia, polyps, malignancy or myomas.
* Women with any cause of pelvic pain as pelvic inflammatory diseases, endometriosis or adenomyosis.
* Women with history of classic upper segment cesarean section or hysterotomy.
* Women with history of previous uterine scars rather than cesarean sections as myomectomy.
* Women with bleeding tendency disorders, taking anticoagulants or having chronic medical conditions as liver diseases, or coagulopathies.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women in child bearing age with history of previous cesarean section and at least 6 months postpartum.
Enrollment: 86 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
correlation between position of the uterus and large Cesarean Scar defect (CSD) | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), which will be correlated to the presence of Large CSD (ratio between the depth (mm) and adjacent myometrial thickness (mm) more than or equal to 0.50)

SECONDARY OUTCOMES:
correlation between position of uterus and Residual myometrial thickness | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), and measuring the thickness of the myometrium over the SCD (mm)
correlation between position of uterus and Depth, Length, Width of SCD | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), and measure depth (mm) and width (mm) of the Cesarean scar defect, while in transverse plane of the uterus measure length (mm) of the cesarean scar defect.
correlation between position of uterus and postmenstrual spotting | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), and correlates to the presence of more than or equal to 2 days of intermenstrual spotting or more than or equal to 2 days of brownish discharge after the end of menstruation if bleeding duration exceeds 7 days (discharge is considered normal if bleeding duration is less than 7 days)
correlation between position of uterus and Abnormal Uterine Bleeding (AUB) | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), and correlates to the presence of AUB as per Figo guideline as regards frequency (in days), duration (in days), regularity (Regular/irregular) and intermenstrual bleeding
correlation between position of uterus and Pelvic Pain | through study completion, up to 6 months
  By using transvaginal ultrasound, the uterus will be examined in a mid sagittal plane to evaluate the position of the uterus that will be described as (Anteverted: the uterus tilts forward at the cervix/ Retroverted: the uterus tilts backward at the cervix), and correlates it to the presence of Dysmenorrhea, Chronic pelvic pain or dyspareunia.
correlation between position of uterus and secondary infertility | through study completion, up to 6 months
  secondary infertility is defined as inability of a couple to conceive after 1 year of regular, unprotected intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: Maya M. Abdelrazek, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt